CLINICAL TRIAL: NCT01512225
Title: Enhancing Breast Milk Production With Domperidone in Mothers of Preterm Neonates
Acronym: EMPOWER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 232-2011
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Low Milk Supply
Keywords: breastmilk; domperidone; preterm
MeSH Terms: conditions — Premature Birth | interventions — Domperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Domperidone for days 1 to 28 (Experimental): Domperidone maleate tablets 10 mg orally three times daily from days 1 to 28
  Interventions: Drug: Domperidone maleate
- Placebo for days 1 to 14 and domperidone for day 15-28 (Placebo Comparator): Identical placebo tablets 10 mg orally three times daily from days 1 to 14 followed by Domperidone maleate tablets 10 mg orally three times daily from days 15 to 28
  Interventions: Drug: Placebo Tablet; Drug: Domperidone maleate

INTERVENTIONS:
Drug: Domperidone maleate — domperidone maleate tablet 10 mg orally three times daily for 28 days
  Arms: Domperidone for days 1 to 28
Drug: Placebo Tablet — placebo tablet 10 mg orally three times daily for 14 days
  Arms: Placebo for days 1 to 14 and domperidone for day 15-28
Drug: Domperidone maleate — domperidone maleate tablet 10 mg orally three times daily for 14 days
  Arms: Placebo for days 1 to 14 and domperidone for day 15-28

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Domperidone in those mothers who are identified as having difficulty with breast milk production to meet the nutritional needs of their infant in the neonatal intensive are unit hospitalization setting, and to determine how it should be considered in the care of mothers and their preterm infants without causing undesirable effects to either the mother or infant.

DETAILED DESCRIPTION:
It is widely acknowledged that recent perinatal and neonatal technological advances (eg. assisted ventilation, surfactant, antenatal corticosteroids) have greatly enhanced the survival rate of very low birth weight and extremely low birth weight infants. A compelling body of evidence now exists to suggest that use of breast milk to feed preterm infants during initial hospitalization positively impacts their neurodevelopment during early childhood and beyond. In order to provide breastmilk, mothers of preterm infants have to begin to produce and mechanically express milk. However, these mothers are often faced with challenges in maintaining an adequate volume that will meet their infants' nutritional needs, as well as declines in production after several weeks despite a myriad of measures designed to assist in production. The primary hypothesis for this study is that Domperidone, through its pharmacologic action on increasing prolactin levels, will assist mothers experiencing inadequate breast milk production in increasing breast milk volumes to a level identified as being sufficient for continued pumping in the hospitalization period.

ELIGIBILITY:
Inclusion Criteria:

* mothers of a preterm infant born < 30 completed weeks gestation (23 0/7-29 6/7 weeks)
* postpartum period of 7-21 days
* mechanically pumping a minimum average of 6 times a day in the 4-7 days prior to enrollment
* experiencing inadequate milk supply defined as providing < 100% of the average of the daily nutritional intake during the previous 72-hour period prior to enrollment based on a fluid intake of 250 mL/kg/d or experiencing a clinical reduction of approximately 20% from a peak volume during the previous 72-hour period prior to enrollment

Exclusion Criteria:

* history of known or suspected cardiac dysrhythmias (tachyarrhythmia, Q-Tc prolongation) or currently on an anti-arrhythmic medication
* currently experiencing mastitis
* previous breast surgery, including augmentation or reduction, nipple piercing and/or the use of nipple rings/studs within the last year, or any reduction
* known chronic or debilitating illness, known abnormal liver function or gastric abnormalities gastrointestinal that will be exacerbated by the use of a prokinetic, examples include hemorrhage or blockage, actively treated with acid reflux which requires treatment for greater than 5 days and includes H2 blockers (occasional use of H2 blockers for heartburn or mild acid reflux is not considered an exclusion) and HIV
* known to have a prolactin-releasing pituitary tumor
* receiving medications known to alter the metabolism and pharmacokinetics of domperidone (eg. oral "azole" antifungals, erythromycin antibiotics, monoamine oxidase inhibitors (MAO) inhibitors) or medications that have dopaminergic or antidopaminergic activity or affect prolactin levels
* mothers of higher order pregnancies (triplet, or more)
* currently smoking 6 or more cigarette per day as reported by the mother

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-05; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth V Asztalos, MD, Principal Investigator — Sunnybrook Research Institute; Marsha Campbell-Yeo, PhD, Principal Investigator — IWK Health Centre; Orlando Da Silva, MD, Principal Investigator — Children's Hospital, London Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asztalos EV, Campbell-Yeo M, da Silva OP, Ito S, Kiss A, Knoppert D; EMPOWER Study Collaborative Group. Enhancing Human Milk Production With Domperidone in Mothers of Preterm Infants. J Hum Lact. 2017 Feb;33(1):181-187. doi: 10.1177/0890334416680176. Epub 2017 Jan 20. PMID 28107101
- [Derived] Asztalos EV, Kiss A, daSilva OP, Campbell-Yeo M, Ito S, Knoppert D; EMPOWER Study Collaborative Group. Role of days postdelivery on breast milk production: a secondary analysis from the EMPOWER trial. Int Breastfeed J. 2019 Jun 4;14:21. doi: 10.1186/s13006-019-0215-z. eCollection 2019. PMID 31171928
- [Derived] Asztalos EV, Kiss A, daSilva OP, Campbell-Yeo M, Ito S, Knoppert D; <italic>EMPOWER</italic> Study Collaborative Group. Evaluating the Effect of a 14-Day Course of Domperidone on Breast Milk Production: A Per-Protocol Analysis from the EMPOWER Trial. Breastfeed Med. 2019 Mar;14(2):102-107. doi: 10.1089/bfm.2018.0175. Epub 2018 Dec 13. PMID 30543461
- [Derived] Asztalos EV, Kiss A, da Silva OP, Campbell-Yeo M, Ito S, Knoppert D; EMPOWER Study Collaborative Group. Pregnancy gestation at delivery and breast milk production: a secondary analysis from the EMPOWER trial. Matern Health Neonatol Perinatol. 2018 Nov 5;4:21. doi: 10.1186/s40748-018-0089-x. eCollection 2018. PMID 30410781
- [Derived] Asztalos EV, Campbell-Yeo M, daSilva OP, Kiss A, Knoppert DC, Ito S. Enhancing breast milk production with Domperidone in mothers of preterm neonates (EMPOWER trial). BMC Pregnancy Childbirth. 2012 Aug 31;12:87. doi: 10.1186/1471-2393-12-87. PMID 22935052

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from June 1, 2012 to June 30, 2015 in 8 Neonatal Intensive Care Units in Canada
Pre-assignment Details: Mothers could be identified in the NICU as early as day 4 until day 18 post-delivery. Additional counseling and support by the lactation consultant with respect to non-pharmacologic techniques were offered. If there was no response to the techniques, the mother was considered eligible for the trial.
Groups:
- Group A: Domperidone: Domperidone 10 mg orally three times daily for 28 days
  Domperidone maleate: domperidone 10 mg orally three times daily for 28 days
- Group B: Placebo + Domperidone: Identical placebo 10 mg orally three times daily for 14 days followed by domperidone 10 mg orally three times daily for 14 days
  Domperidone maleate plus placebo: identical placebo 10 mg orally three times daily for 14 days followed by domperidone 10 mg orally three times daily for 14 days
Period: Overall Study
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Started | 45 | 45
Provided Day 14 Volume | 45 | 40
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Full Range); unit: years] | 31.25 [20.96 to 40.59] | 33.56 [23.23 to 39.50] | 32.41 [20.96 to 40.59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity was self-declared
  Participants
    Caucasian | 29 | 30 | 59
    Black | 6 | 4 | 10
    Asian | 8 | 8 | 16
    Aboriginal | 0 | 1 | 1
    Other | 2 | 2 | 4
Parity [Count of Participants; unit: Participants]
  0 | 28 | 33 | 61
  >/= 1 | 17 | 12 | 29
Type of pregnancy [Count of Participants; unit: Participants]
  Singleton | 38 | 39 | 77
  Twins | 7 | 6 | 13
Mean milk Volume at entry [Mean (Standard Deviation); unit: millilitres] | 121 (96) | 115 (95) | 118 (96)

OUTCOME MEASURES:

1. Primary Outcome: Increase in Breast Milk Production
Description: The primary outcome is the difference in the proportion of women having a 50% increase in breast milk volume at the end of 14 days of treatment with domperidone compared to mothers receiving placebo (mean day 14 volume minus mean day 0 volume at entry).
Time Frame: Day 0 to day 14
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Domperidone: Domperidone 10 mg orally three times daily for 28 days
- Group B: Placebo + Domperidone: Identical placebo 10 mg orally three times daily for 14 days followed by domperidone 10 mg orally three times daily for 14 days
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Number analyzed (Participants) | 45 | 45
Participants | 35 | 26

2. Secondary Outcome: Increase in Breast Milk Volume on Day 28
Description: Number of mothers who achieved 50% increase in milk volume on day 28
Time Frame: day 0 to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Number analyzed (Participants) | 45 | 45
Participants | 31 | 28

3. Secondary Outcome: Mean Breast Milk Volumes on Day 14
Description: Mean milk volumes between the two groups at 14 days of study intervention
Time Frame: Day 0 and day 14
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Number analyzed (Participants) | 45 | 45
millilitres | 267 (189) | 217 (168)

4. Secondary Outcome: Mean Breast Milk Volumes on Day 28
Description: Mean milk volumes between the two groups at 28 days of study intervention
Time Frame: day 0 and 28
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Number analyzed (Participants) | 45 | 45
millilitres | 290 (211) | 302 (230)

5. Secondary Outcome: Mean Volume Change From Day 0 to Day 14
Description: change on the volume of milk from day 0 to day 14 between the two groups
Time Frame: days 0 and 14
Measure: Mean (Full Range); unit: millilitres
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Number analyzed (Participants) | 45 | 45
millilitres | 254 [-100 to 2129] | 175 [-100 to 923]

6. Secondary Outcome: Mean Volume Change on the Volume of Milk From Day 15 to Day 28
Description: change on the volume of milk from day 15 to day 28 between the two groups
Time Frame: day 15 and day 28
Measure: Mean (Full Range); unit: millilitres
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Number analyzed (Participants) | 45 | 45
millilitres | 22 [-68 to 200] | 49 [-100 to 254]

7. Secondary Outcome: Provision of Breast Milk at Term Gestation
Description: provision of breast milk as the primary source of nutrition
Time Frame: term gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Number analyzed (Participants) | 45 | 45
Participants | 26 | 27

8. Secondary Outcome: Provision of Breast Milk at 6 Weeks Post Term Gestation
Description: Provision of breast milk at 6 weeks post term gestation as primary source of nutrition
Time Frame: 6 weeks post term gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Number analyzed (Participants) | 45 | 45
Participants | 19 | 20

ADVERSE EVENTS:
Arm/Group | Group A: Domperidone | Group B: Placebo + Domperidone
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 10/45 | 3/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Domperidone (N=45) | Group B: Placebo + Domperidone (N=45)
Headache (Nervous system disorders) | 10 (31) | 3 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No